CLINICAL TRIAL: NCT05447143
Title: Examination of the Effect of Home Exercise Program on Various Parameters in Patients With Multiple Sclerosis: A Randomized Controlled Single-Blind Trial
Brief Title: Effect of Home Exercise Program on Various Parameters in Patients With Multiple Sclerosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Muğla Sıtkı Koçman University (Other)
Responsible Party: Principal Investigator, Banu BAYAR, Principal investigator, Head of Physiotherapy and Rehabilitation Department, Pt. PhD. Prof., Muğla Sıtkı Koçman University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 200301
Record Dates: First submitted 2022-07-03; First posted 2022-07-07 (Actual); Last update posted 2022-07-20 (Actual); Status verified 2022-07

CONDITIONS: Multiple Sclerosis; Exercise Program; Telerehabilitation; Autoimmune Disorder
Keywords: MS (Multiple Sclerosis); Exercise, Physical; Exercise Therapy; Physical Exertion
MeSH Terms: conditions — Multiple Sclerosis; Autoimmune Diseases; Motor Activity

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control Group (CG) (Other): The control group will be queued to be included in the exercise program and participants' routine treatment will continue.
  Interventions: Other: Fatigue Severity Scale; Other: Berg Balance Test; Other: Time up and go- 25 steps walking test; Other: Multiple Sclerosis Quality of Life; Other: Brief International Cognitive Assessment for MS (BICAMS); Other: Beck Depression and Anxiety Scale
- Video Group (VG) (Experimental): The exercise will be given as a video and participants will be asked to continue the exercises for 8 weeks, 3 days a week. Patients will be contacted by phone every week to ask if participants have any problems with the exercise program and their compliance.
  Interventions: Other: Fatigue Severity Scale; Other: Berg Balance Test; Other: Time up and go- 25 steps walking test; Other: Multiple Sclerosis Quality of Life; Other: Brief International Cognitive Assessment for MS (BICAMS); Other: Beck Depression and Anxiety Scale
- Brochure Group (BG) (Experimental): Exercise will be given as a brochure and participants will be asked to continue the exercises given for 8 weeks, 3 days a week. Visual feedback will be provided by asking participants to mark the exercise tracking chart on the exercise brochures.
  Interventions: Other: Fatigue Severity Scale; Other: Berg Balance Test; Other: Time up and go- 25 steps walking test; Other: Multiple Sclerosis Quality of Life; Other: Brief International Cognitive Assessment for MS (BICAMS); Other: Beck Depression and Anxiety Scale

INTERVENTIONS:
Other: Fatigue Severity Scale — Evaluation for severity of fatigue
Other: Berg Balance Test — Evaluation of balance
Other: Time up and go- 25 steps walking test — Evaluation for walking
Other: Multiple Sclerosis Quality of Life — Evaluation of quality of life
Other: Brief International Cognitive Assessment for MS (BICAMS) — Evaluation of cognitive functions
Other: Beck Depression and Anxiety Scale — Evaluation of depression and anxiety

SUMMARY:
Multiple Sclerosis (MS) is a chronic, inflammatory, neurodegenerative, and autoimmune disease that progresses with progressive neurological dysfunction and affects the central nervous system. A multidisciplinary rehabilitation approach is crucial in the systematic and supportive treatment of MS. Exercise training is a therapeutic approach that minimizes functional capacity loss and slows progression in MS. Randomized controlled studies have shown that exercise training improves physical fitness, reduces motor fatigue, and improves the quality of life and psychological state in individuals with MS.

When the literature is examined, it is seen that popular exercises such as pilates, yoga, and Tai-Chi are used in addition to aerobics, strengthening, endurance, and stretching exercises in the treatment of individuals with MS. In order to eliminate the economic burden, which is one of the exercise barriers of individuals, and to gain exercise habits, home exercise programs should be expanded. When the literature is examined, it is emphasized that the importance of home exercise programs is emphasized, and it is very important in the treatment of patients who cannot attend an exercise program, especially by going to any center for various reasons. However, there is little information on the effectiveness and content of home exercise programs in patients with MS. From this point of view, this study is capable of supporting the missing part of the literature.

ELIGIBILITY:
Inclusion Criteria:

1. To be between the ages of 18-65
2. Being diagnosed with MS according to McDonald criteria
3. Having an EDSS score between 0-5.5
4. Being in the Relapsing Remitting class as a clinical subtype of MS
5. Not having any nervous system pathology other than MS
6. Not having an MS attack in the last 1 month
7. To ensure full cooperation and adaptation throughout the study.

Exclusion Criteria:

1. Being in an exacerbation period
2. To have participated in a regular physical activity program in the last 6 months
3. Having an orthopedic, cardiopulmonary or psychiatric disease that prevents exercise
4. Continuing another exercise therapy
5. Not volunteering to participate in the study
6. Having problems with reading comprehension

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2021-09-30 (Actual); Primary Completion 2021-11-30 (Actual); Study Completion 2022-06-15 (Actual)

PRIMARY OUTCOMES:
Timed up and go with 25 steps walking test | Baseline- after 8 weeks (after treatment)
  Timed up and go: Patients wear their regular footwear and can use a walking aid, if needed.
  1. The patient starts in a seated position
  2. The patient stands up upon therapist's command: walks 3 meters, turns around, walks back to the chair and sits down.
  3. The time stops when the patient is seated.
  4. Be sure to document the assistive device used. Note: A practice trial should be completed before the timed trial. High falling risk>13.5 seconds.
  The 25 steps walking test is a quantitative mobility and leg function performance test based on a timed 25-walk. The patient is directed to one end of a clearly marked 25-foot course and is instructed to walk 25 feet as quickly as possible, but safely. The time is recorded.
Fatigue Severity Scale | Baseline- after 8 weeks (after treatment)
  The Fatigue Severity Scale questionnaire contains nine statements that rate the severity of fatigue symptoms. A total score of less than 36 suggests that patient may not be suffering from fatigue. A higher score is indicated high level of fatigue.
Brief International Cognitive Assessment for MS (BICAMS) | Baseline- after 8 weeks (after treatment)
  The Brief International Cognitive Assessment for MS (BICAMS) initiative was undertaken to recommend a brief, cognitive assessment for MS that is optimized for small centers. BICAMS was particularly focused on international use, to facilitate comparison across settings. An expert committee of twelve neurologists and neuropsychologists representing the main cultural groups that have so far contributed extensive data about cognitive dysfunction in MS was convened. The opinions generated from the meeting are published elsewhere. Consensus was also achieved on optimal measures for learning and memory in MS patients, time permitting: the initial learning trials of the second edition of the California Verbal Learning Test (CVLT2) and the revised Brief Visuospatial Memory Test (BVMTR).
Berg Balance Scale | Baseline- after 8 weeks (after treatment)
  The Berg Balance Scale (BBS) is used to objectively determine a patient's ability (or inability) to safely balance during a series of predetermined tasks. It is a 14 item list with each item consisting of a five-point ordinal scale ranging from 0 to 4, with 0 indicating the lowest level of function and 4 the highest level of function and takes approximately 20 minutes to complete. A score of 56 indicates functional balance.
  A score of < 45 indicates individuals may be at greater risk of falling.

SECONDARY OUTCOMES:
Beck Depression and Anxiety Scale | Baseline- after 8 weeks (after treatment)
  The Beck Depression Scale is a 21-item self-reported questionnaire in which each item consists of four statements indicating different levels of severity of a particular symptom experienced over the past week. Scores for all 21 items are summed up to yield a single depression score. Scores of 0-12 are considered in the normal range, 13-18 as mild, 19-28 as moderate, and scores of 29-63 are considered to indicate severe depression.
  The Beck Anxiety Scale consists of 21 symptoms that are rated on a four-point severity scale referring to the experience of symptoms over the past week. Scores for the 21 items are summed up to yield a single anxiety score. Scores between 0 and 17 are considered as normal and mild anxiety, whereas scores over 25 are considered as severe anxiety.
Mulitple Sclerosis Quality of life- 54 | Baseline- after 8 weeks (after treatment)
  The MSQOL-54 is a multidimensional health-related quality of life measure that combines both generic and MS-specific items into a single instrument. The developers utilized the SF-36 as the generic component to which 18 items were added to tap MS-specific issues such as fatigue, cognitive function, etc. This 54-item instrument generates 12 subscales along with two summary scores, and two additional single-item measures. The subscales are: physical function, role limitations-physical, role limitations-emotional, pain, emotional well-being, energy, health perceptions, social function, cognitive function, health distress, overall quality of life, and sexual function. The summary scores are the physical health composite summary and the mental health composite summary. The single item measures are satisfaction with sexual function and change in health.

CONTACTS AND LOCATIONS:
Locations (1):
- Muğla Sıtkı Koçman University, Muğla, Merkez, Turkey (Türkiye)